CLINICAL TRIAL: NCT03504540
Title: Comparison of Complement Factors and Genetic Polymorphisms of AMD Between Patients With Systemic Lupus Erythematosus (SLE) With and Without Retinal "Pseudo-drusen-like" Deposits: Case-control Study (PLAMD)
Brief Title: Comparison of Complement Factors and Genetic Polymorphisms of AMD Between Patients With Systemic Lupus Erythematosus (SLE) With and Without Retinal "Pseudo-drusen-like" Deposits: Case-control Study (PL-AMD)
Acronym: PL-AMD
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2018_1
Record Dates: First submitted 2018-04-06; First posted 2018-04-20 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Lupus Erythematosus; Lupus Erythematosus, Systemic; Age Related Macular Degeneration
Keywords: Lupus Erythematosus, Systemic; Age Related Macular Degeneration; "Pseudo-drusen-like" deposits
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Macular Degeneration | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case (with pseudo-drusen-like deposits): Patients with lupus, treated or not with antimalarial drugs, with "pseudo-drusen-like" deposits
  Interventions: Procedure: Blood test
- Control (without pseudo-drusen-like deposits): Patients with lupus, treated or not with antimalarial drugs, without "pseudo-drusen-like" deposits
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — Blood test for complement factors and genetic polymorphisms of AMD analysis

SUMMARY:
The rationale of this research is to determine if patients with lupus and presenting retinal "pseudo-drusen-like" deposits have genetic and complement-related similarities with AMD patients.

Based on the results obtained, this study could lead to future research that could better target the treatment of patients with lupus or patients with AMD (Age related Macular Degeneration).

The primary objective is to check if patients with lupus, treated or not with antimalarial drugs, with "pseudo-drusen-like" deposits have a different complement profile (functional exploration of complement, complement factors, genetic complement polymorphisms involved in AMD) compared to patients without "pseudo-drusen-like" deposits.

ELIGIBILITY:
Inclusion Criteria:

* Systemic lupus erythematosus
* Case patients : with "pseudo-drusen-like" deposit
* Control patients : without "pseudo-drusen-like" deposit

Exclusion Criteria:

* Patient under a measure of legal protection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with lupus, treated or not with APS, with ou without "pseudo-drusen-like" deposits
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Comparison of AMD genetic polymorphisms between case and control patients | Baseline
Comparison of complement factors between case and control patients | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation ophtalmologique Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided